CLINICAL TRIAL: NCT03590613
Title: A Single-centre, Randomized, Double-blind, Dose-ascending, Placebo-controlled Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Oral TID Doses (One Day) of GSK2982772 in Japanese Healthy Male Subjects
Brief Title: Phase I Study of GSK2982772 in Japanese Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 205037
Record Dates: First submitted 2018-07-06; First posted 2018-07-18 (Actual); Results first posted 2019-09-17 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-09

CONDITIONS: Autoimmune Diseases
Keywords: Sentinel-dosing; GSK2982772; Japnese; Dose-ascending; Crossover; Healthy
MeSH Terms: conditions — Autoimmune Diseases | interventions — GSK2982772

STUDY DESIGN:
Intervention Model Description: Study will comprise of four TPs, each of at least 7 days in duration with subjects in-house for 4 nights (through 72 hours after the first dose). During each TP, subjects will be admitted to the unit, day before dosing and will be discharged after completion of 72 hours post-dose assessments. dose will be administered TID, in an ascending manner. Every individual subject will receive placebo and GSK2982772 (60, 120,240 mg TID) as per assigned sequence. For TID dosing, GSK2982772 or placebo will be administered at 0 hour (the first dosing), 7 hour (the second dosing) and 14 hour (the third dosing) on Day 1 in each period. On Day 1, subjects will fast 8hour overnight prior to first dose. breakfast will be served approximately 2hour after first dose. Lunch and dinner will be served between 2 to 3hour prior to second and third doses, respectively. A washout of atleast 7-days between the TP doses for each individual subject.
Who Masked: Participant, Care Provider, Investigator
Masking Description: It is a double-blinded study, where the subjects, investigators and the site-staff will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sequence 1: Placebo TID then 60 TID then 120 TID then 240 TID (Experimental): The eligible subjects in this arm will receive placebo TID in TP1, GSK2982772 60 mg TID in TP2, GSK2982772 120mg TID in TP3 and GSK2982772 240 mg TID in TP4. GSK2982772 or placebo will be administered at 0 hour (the first dosing), 7 hours (the second dosing) and 14 hours (the third dosing) on Day 1 in each TP. Subjects will fast overnight for 8 hours before first dose. Each TP will be followed by a washout period of at least 7 days, for each subject.
  Interventions: Drug: GSK2982772; Drug: Placebo
- Sequence 2: 60 TID then Placebo TID then 120 TID then 240 TID (Experimental): The eligible subjects in this arm will receive GSK2982772 60 mg TID in TP1, placebo TID in TP2, GSK2982772 120mg TID in TP3 and GSK2982772 240 mg TID in TP4. GSK2982772 or placebo will be administered at 0 hour (the first dosing), 7 hours (the second dosing) and 14 hours (the third dosing) on Day 1 in each TP. Subjects will fast overnight for 8 hours before first dose. Each TP will be followed by a washout period of at least 7 days, for each subject.
  Interventions: Drug: GSK2982772; Drug: Placebo
- Sequence 3: 60 TID then 120 TID then Placebo TID then 240 TID (Experimental): The eligible subjects in this arm will receive GSK2982772 60 mg TID in TP1, GSK2982772 120mg TID in TP2, placebo TID in TP3 and GSK2982772 240 mg TID in TP4. GSK2982772 or placebo will be administered at 0 hour (the first dosing), 7 hours (the second dosing) and 14 hours (the third dosing) on Day 1 in each TP. Subjects will fast overnight for 8 hours before first dose. Each TP will be followed by a washout period of at least 7 days, for each subject.
  Interventions: Drug: GSK2982772; Drug: Placebo
- Sequence 4: 60 TID then 120 TID then 240 TID then Placebo TID (Experimental): The eligible subjects in this arm will receive GSK2982772 60 mg TID in TP1, GSK2982772 120mg TID in TP2, GSK2982772 240 mg TID in TP3 and placebo TID in TP4. GSK2982772 or placebo will be administered at 0 hour (the first dosing), 7 hours (the second dosing) and 14 hours (the third dosing) on Day 1 in each TP. Subjects will fast overnight for 8 hours before first dose. Each TP will be followed by a washout period of at least 7 days, for each subject.
  Interventions: Drug: GSK2982772; Drug: Placebo

INTERVENTIONS:
Drug: GSK2982772 — GSK2982772 will be available as white to almost white, round, film coated tablets to be administered via oral route
Drug: Placebo — Placebo matching GSK2982772 will be available as white to almost white, round, film coated tablets to be administered via oral route.

SUMMARY:
The study plans to enroll approximately 12 subjects. The main objective of the study is to assess the safety, tolerability and pharmacokinetics (PK) of the three times a day (TID), dosing of GSK2982772, in Japanese healthy male subjects. The study will comprise of four study periods each at least 7 days in duration with subjects in-house for 4 nights (through 72 hrs after the first dose). During each treatment period (TP), subjects will be admitted to the unit the day before dosing and will be discharged after completion of the 72 hours post-dose assessments. There will be a washout of atleast 7-days between the TP doses for each individual, post which there will be 7-days follow-up. The dose range proposed in this study is based on a low starting dose, which will be escalated to the highest dose that is intended for the Phase 2b dose range study. The decision to proceed to the next dose-level, of GSK2982772 within the study will be made by principal investigator and GSK Medical Monitor per each dosing periods. The study duration is approximately 22 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be 20 to 64 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by the Investigators based on a medical evaluation including medical history, physical examination, neurological examination, laboratory tests, and ECG. A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the Investigators in consultation with the GSK Medical Monitor agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Body weight >= 50 kilogram (kg) and body mass index (BMI) within the range 18.5-24.9 kg/meter square (inclusive).
* Japanese male subjects must agree to use contraception as detailed in protocol during the treatment period and until follow up visit.
* Capable of giving informed consent as described in the protocol.

Exclusion Criteria:

* History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study treatment; or interfering with the interpretation of data.
* Abnormal blood pressure as determined by the investigators.
* Symptomatic herpes zoster within 3 months prior to screening.
* Evidence of active or latent Tuberculosis (TB) as documented by medical history and examination, chest X-rays (anterior and lateral), and TB testing (T Spot. TB)
* ALT >1.5 times upper limit of normal (ULN).
* Bilirubin >1.5 times ULN (isolated bilirubin >1.5 times ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%)
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* History of active infections within 14 days of first receiving study medication.
* Corrected Q-T interval (QTc) obtained using the Fridericia's formula (QTcF) > 450 millisecond.
* History or diagnosis of obstructive sleep apnoea, or a significant respiratory disorder. Childhood asthma that was fully resolved is permitted.
* History of active Suicidal Ideation Behavior within the past 6 months or any history of attempted suicide in a subject's lifetime.
* History or current evidence of febrile seizures, epilepsy, convulsions, significant head injury, or other significant neurologic conditions.
* Past or intended use of over-the-counter or prescription medication including herbal medications within 14 days prior to dosing; live vaccine(s) within 1 month prior to screening, or plans to receive such vaccines during the study.
* History of donation of blood or blood products >= 400 mL within 3 months or >= 200 mL within 1 month prior to screening.
* Exposure to more than 4 new chemical entities within 12 months prior to the first dosing day.
* The subject has participated in a other clinical study or other medical research within 4 months prior to the first dosing day in the current study.
* Subject is positive Serological test for syphilis Rapid Plasma Reagin [RPR] and Treponema pallidum [TP]), Tuberculosis, human immunodeficiency virus (HIV) Antigen/Antibody, Hepatitis B surface antigen (HbsAg), Hepatitis C virus (HCV) antibody, or Human T-cell leukemia virus type 1 (HTLV-1) antibody at screening.
* Positive pre-study drug screen.
* Regular use of known drugs of abuse.
* Regular alcohol consumption within 6 months prior to the study defined as: for an average weekly intake of > 14 units for males. One unit is equivalent to 350 mL of beer, 150 mL of wine or 45 mL of 80 proof distilled spirits.
* Smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* Sensitivity to any of the study treatments, or components thereof, or drug or other allergy that, in the opinion of the investigators or GSK Medical Monitor, contraindicates participation in the study.

Ages: 20 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 13 (Actual)
Dates: Start 2018-07-19 (Actual); Primary Completion 2018-09-21 (Actual); Study Completion 2018-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Fukuoka, Japan

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD is made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency

REFERENCES:
- [Derived] Tompson DJ, Davies C, Scott NE, Cannons EP, Kostapanos M, Gross AS, Powell M, Ino H, Shimamura R, Ogura H, Nagakubo T, Igarashi H, Nakano A. Comparison of the Pharmacokinetics of RIPK1 Inhibitor GSK2982772 in Healthy Western and Japanese Subjects. Eur J Drug Metab Pharmacokinet. 2021 Jan;46(1):71-83. doi: 10.1007/s13318-020-00652-2. PMID 33165774

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a 4-way crossover, single-center, randomized, double-blind, dose-ascending, placebo (PBO)-controlled study to evaluate the safety, tolerability, and pharmacokinetics of oral TID doses (thrice a day) of GSK2982772 in healthy male Japanese participants
Pre-assignment Details: A total of 13 healthy male Japanese participants were enrolled in the study to receive GSK2982772 and PBO from a single center in Japan
Groups:
- Treatment Sequence A: PBO TID /60mg TID /120mg TID /240mg TID: Participants in this arm received PBO TID in treatment period (TP) 1, GSK2982772 60 milligram (mg) TID in TP2, GSK2982772 120 mg TID in TP3 and GSK2982772 240 mg TID in TP4. GSK2982772 and placebo was administered at 0 hour (starting dose), 7 hours (second dose) and 14 hours (third dose) on Day 1 in each TP. Participants had fasted overnight for 8 hours before first dose. Each TP was followed by a washout period of at least 7 days, for each participant.
- Treatment Sequence B: 60mg TID /PBO TID /120mg TID /240mg TID: Participants in this arm received GSK2982772 60 mg TID in TP1, PBO TID in TP2, GSK2982772 120mg TID in TP3 and GSK2982772 240 mg TID in TP4. GSK2982772 and placebo was administered at 0 hour (starting dose), 7 hours (second dose) and 14 hours (third dose) on Day 1 in each TP. Participants had fasted overnight for 8 hours before first dose. Each TP was followed by a washout period of at least 7 days, for each participant.
- Treatment Sequence C: 60mg TID/ 120mg TID/ PBO TID/ 240mg TID: Participants in this arm received GSK2982772 60 mg TID in TP1, GSK2982772 120mg TID in TP2, PBO TID in TP3 and GSK2982772 240 mg TID in TP4. GSK2982772 and placebo was administered at 0 hour (starting dose), 7 hours (second dose) and 14 hours (third dose) on Day 1 in each TP. Participants had fasted overnight for 8 hours before first dose. Each TP was followed by a washout period of at least 7 days, for each participant.
- Treatment Sequence D: 60mg TID /120mg TID /240mg TID /PBO TID: Participants in this arm received GSK2982772 60 mg TID in TP1, GSK2982772 120mg TID in TP2, GSK2982772 240 mg TID in TP3 and PBO TID in TP4. GSK2982772 and placebo was administered at 0 hour (starting dose), 7 hours (second dose) and 14 hours (third dose) on Day 1 in each TP. Participants had fasted overnight for 8 hours before first dose. Each TP was followed by a washout period of at least 7 days, for each participant.
Period: Period 1, 4 Days
Arm/Group | Treatment Sequence A: PBO TID /60mg TID /120mg TID /240mg TID | Treatment Sequence B: 60mg TID /PBO TID /120mg TID /240mg TID | Treatment Sequence C: 60mg TID/ 120mg TID/ PBO TID/ 240mg TID | Treatment Sequence D: 60mg TID /120mg TID /240mg TID /PBO TID
Started | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0
Period: Period 1, Wash-out, at Least 3 Days
Arm/Group | Treatment Sequence A: PBO TID /60mg TID /120mg TID /240mg TID | Treatment Sequence B: 60mg TID /PBO TID /120mg TID /240mg TID | Treatment Sequence C: 60mg TID/ 120mg TID/ PBO TID/ 240mg TID | Treatment Sequence D: 60mg TID /120mg TID /240mg TID /PBO TID
Started | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0
Period: Period 2, 4 Days
Arm/Group | Treatment Sequence A: PBO TID /60mg TID /120mg TID /240mg TID | Treatment Sequence B: 60mg TID /PBO TID /120mg TID /240mg TID | Treatment Sequence C: 60mg TID/ 120mg TID/ PBO TID/ 240mg TID | Treatment Sequence D: 60mg TID /120mg TID /240mg TID /PBO TID
Started | 3 | 3 | 3 | 4 (One additional participant was enrolled in Period 2.)
Completed | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 1
Period: Period 2, Wash-out, at Least 3 Days
Arm/Group | Treatment Sequence A: PBO TID /60mg TID /120mg TID /240mg TID | Treatment Sequence B: 60mg TID /PBO TID /120mg TID /240mg TID | Treatment Sequence C: 60mg TID/ 120mg TID/ PBO TID/ 240mg TID | Treatment Sequence D: 60mg TID /120mg TID /240mg TID /PBO TID
Started | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0
Period: Period 3, 4 Days
Arm/Group | Treatment Sequence A: PBO TID /60mg TID /120mg TID /240mg TID | Treatment Sequence B: 60mg TID /PBO TID /120mg TID /240mg TID | Treatment Sequence C: 60mg TID/ 120mg TID/ PBO TID/ 240mg TID | Treatment Sequence D: 60mg TID /120mg TID /240mg TID /PBO TID
Started | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0
Period: Period 3,Wash-out, at Least 3 Days
Arm/Group | Treatment Sequence A: PBO TID /60mg TID /120mg TID /240mg TID | Treatment Sequence B: 60mg TID /PBO TID /120mg TID /240mg TID | Treatment Sequence C: 60mg TID/ 120mg TID/ PBO TID/ 240mg TID | Treatment Sequence D: 60mg TID /120mg TID /240mg TID /PBO TID
Started | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0
Period: Period 4, 4 Days
Arm/Group | Treatment Sequence A: PBO TID /60mg TID /120mg TID /240mg TID | Treatment Sequence B: 60mg TID /PBO TID /120mg TID /240mg TID | Treatment Sequence C: 60mg TID/ 120mg TID/ PBO TID/ 240mg TID | Treatment Sequence D: 60mg TID /120mg TID /240mg TID /PBO TID
Started | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All study participants received GSK2982772 and PBO in four treatment sequences (A,B,C &D) at 0 hour (starting dose), 7 hours (second dose) and 14 hours (third dose) on Day 1 in each TP.
Arm/Group | All Study Participants
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: Years] | 26.2 (7.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 13
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian-Japanese/East Asian/South East AsianHeritage | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. A SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect, associated with liver injury and impaired liver function or any other situations as per medical or scientific judgement. Safety population comprised of all participants who have received at least one dose of study treatment. This population was used for the safety analyses.
Time Frame: From the day of first dose to 39 days
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Participants were administered PBO matching GSK2982772 via oral route using a 7 hours dosing interval in each TP.
- GSK2982772 60 mg: Participants were administered GSK2982772 60 mg via oral route using a 7 hours dosing interval in each TP.
- GSK2982772 120 mg: Participants were administered GSK2982772 120 mg via oral route using a 7 hours dosing interval in each TP.
- GSK2982772 240 mg: Participants were administered GSK2982772 240 mg via oral route using a 7 hours dosing interval in each TP.
Arm/Group | Placebo | GSK2982772 60 mg | GSK2982772 120 mg | GSK2982772 240 mg
Number analyzed (Participants) | 12 | 12 | 12 | 12
Participants
  Any AE | 0 | 1 | 0 | 0
  Any SAE | 0 | 0 | 0 | 0

2. Primary Outcome: Change From Baseline in Clinical Chemistry Parameters
Description: Blood samples were collected for the analysis of clinical chemistry parameters including: glucose, calcium, cholesterol, chloride, high density lipoprotein (HDL) cholesterol, potassium, low density lipoprotein (LDL) cholesterol, phosphate, sodium, triglycerides and urea. Baseline value was the latest pre-dose (Day -1) assessment with a non-missing value, including those from unscheduled visits. Change from Baseline is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day -1) and at 72 hours at each treatment period
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Placebo | GSK2982772 60 mg | GSK2982772 120 mg | GSK2982772 240 mg
Number analyzed (Participants) | 12 | 12 | 12 | 12
Millimoles per liter
  Glucose | -0.240543 (0.1426732) | -0.282176 (0.2348638) | -0.240543 (0.2902134) | -0.226666 (0.2554319)
  Calcium | 0.016633 (0.0683974) | 0.058217 (0.0341987) | -0.022871 (0.0732901) | -0.004158 (0.1036024)
  Cholesterol | 0.000000 (0.2092177) | 0.073270 (0.2657498) | 0.015085 (0.3458001) | -0.049565 (0.3560217)
  Chloride | 1.1 (1.38) | 0.2 (2.25) | 1.2 (1.59) | 0.6 (1.68)
  HDL Cholesterol | -0.071115 (0.1097839) | -0.034480 (0.1070976) | -0.084045 (0.1046815) | -0.116370 (0.0578247)
  Potassium | -0.06 (0.156) | 0.01 (0.329) | 0.03 (0.501) | -0.07 (0.419)
  LDL Cholesterol | 0.036635 (0.1670318) | 0.101285 (0.1673953) | 0.017240 (0.2663211) | -0.043100 (0.1926790)
  Phosphate | 0.064580 (0.0963795) | 0.053817 (0.1210793) | 0.002691 (0.1155721) | 0.018836 (0.1366196)
  Sodium | 1.5 (1.78) | 1.3 (1.72) | 0.9 (1.93) | 1.4 (1.83)
  Triglycerides | 0.19398 (0.117614) | 0.12618 (0.153495) | 0.13372 (0.286674) | 0.13466 (0.368074)
  Urea | -0.09223 (0.656241) | -0.21123 (0.796454) | -0.03273 (0.309530) | -0.31238 (0.705860)

3. Primary Outcome: Change From Baseline in Clinical Chemistry Parameters: Albumin and Protein
Description: Blood samples were collected for the analysis of clinical chemistry parameters including: albumin and protein. Baseline value was the latest pre-dose (Day -1) assessment with a non-missing value, including those from unscheduled visits. Change from Baseline is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day -1) and at 72 hours at each Treatment Period
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Placebo | GSK2982772 60 mg | GSK2982772 120 mg | GSK2982772 240 mg
Number analyzed (Participants) | 12 | 12 | 12 | 12
Grams per liter
  Albumin | -1.4 (2.64) | -0.4 (1.62) | -1.6 (2.47) | -2.5 (3.23)
  Protein | -1.3 (3.96) | 0.8 (2.12) | -2.1 (3.70) | -2.3 (4.27)

4. Primary Outcome: Change From Baseline in Clinical Chemistry Parameters: Alkaline Phosphate (ALP), Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), Creatinine Kinase (CK), Gamma Glutamyl Transferase (GGT) and Lactate Dehydrognase (LDH)
Description: Blood samples were collected for the analysis of clinical chemistry parameters including: ALP, ALT, AST, CK, GGT and LDH. Baseline value was the latest pre-dose (Day -1) assessment with a non-missing value, including those from unscheduled visits. Change from Baseline is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day -1) and at 72 hours at each Treatment Period
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | Placebo | GSK2982772 60 mg | GSK2982772 120 mg | GSK2982772 240 mg
Number analyzed (Participants) | 12 | 12 | 12 | 12
International units per liter
  ALP | -9.1 (17.32) | -6.8 (12.63) | -10.6 (14.41) | -9.0 (14.65)
  ALT | -0.5 (3.66) | 0.5 (2.47) | -2.2 (3.33) | -1.3 (4.59)
  AST | -0.6 (2.68) | 0.3 (1.76) | -1.8 (3.28) | -2.5 (6.64)
  CK | -19.1 (14.95) | -34.2 (21.70) | -51.7 (48.61) | -39.6 (32.91)
  GGT | -0.5 (0.67) | -0.5 (1.62) | -1.8 (2.93) | -1.5 (2.32)
  LDH | -17.7 (9.76) | -11.3 (8.01) | -21.6 (14.92) | -21.3 (10.34)

5. Primary Outcome: Change From Baseline in Clinical Chemistry Parameter: Amylase
Description: Blood samples were collected for the analysis of clinical chemistry parameter: amylase. Baseline value was the latest pre-dose (Day -1) assessment with a non-missing value, including those from unscheduled visits. Change from Baseline is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day -1) and at 72 hours at each Treatment Period
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Units per liter
Arm/Group | Placebo | GSK2982772 60 mg | GSK2982772 120 mg | GSK2982772 240 mg
Number analyzed (Participants) | 12 | 12 | 12 | 12
Units per liter | 4.2 (10.56) | 9.1 (6.26) | 4.4 (9.34) | 1.1 (8.40)

6. Primary Outcome: Change From Baseline in Clinical Chemistry Parameters: Direct Bilirubin, Bilirubin, Creatinine and Urate (Uric Acid)
Description: Blood samples were collected for the analysis of clinical chemistry parameters:direct bilirubin, bilirubin, creatinine and urate. Baseline value was the latest pre-dose (Day -1) assessment with a non-missing value, including those from unscheduled visits. Change from Baseline is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day -1) and at 72 hours at each Treatment Period
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Placebo | GSK2982772 60 mg | GSK2982772 120 mg | GSK2982772 240 mg
Number analyzed (Participants) | 12 | 12 | 12 | 12
Micromoles per liter
  Direct bilirubin | 0.428 (1.0629) | 0.285 (0.9873) | 0.143 (1.1432) | -0.285 (0.9873)
  Bilirubin | 2.850 (4.7998) | 2.850 (4.7998) | 1.568 (5.9441) | -0.428 (4.0679)
  Creatinine | 0.8840 (7.47252) | 0.5157 (4.46730) | 0.6630 (5.25184) | 1.6943 (3.97949)
  Urate | 21.8093 (29.82999) | 9.4177 (23.16992) | 17.8440 (17.93389) | 8.4263 (27.95138)

7. Primary Outcome: Change From Baseline in Clinical Chemistry Parameter: C-reactive Protein (CRP) of TID Doses for One Day of GSK2982772
Description: Blood samples were collected for the analysis of clinical chemistry parameter: CRP. Baseline value was the latest pre-dose (Day -1) assessment with a non-missing value, including those from unscheduled visits. Change from Baseline is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day -1) and at 72 hours at each Treatment Period
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Milligrams per liter
Arm/Group | Placebo | GSK2982772 60 mg | GSK2982772 120 mg | GSK2982772 240 mg
Number analyzed (Participants) | 12 | 12 | 12 | 12
Milligrams per liter | -0.078 (0.2290) | -0.016 (0.0268) | -0.050 (0.1028) | 0.126 (0.5390)

8. Primary Outcome: Change From Baseline in Hematology Parameter: Hematocrit
Description: Blood samples were collected for the analysis of hematology parameter: hematocrit. Baseline value was the latest pre-dose (Day -1) assessment with a non-missing value, including those from unscheduled visits. Change from Baseline is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day -1) and at 72 hours at each Treatment Period
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Percentage of red blood cells in blood
Arm/Group | Placebo | GSK2982772 60 mg | GSK2982772 120 mg | GSK2982772 240 mg
Number analyzed (Participants) | 12 | 12 | 12 | 12
Percentage of red blood cells in blood | 0.0039 (0.01946) | 0.0075 (0.01332) | -0.0048 (0.01434) | -0.0043 (0.02172)

9. Primary Outcome: Change From Baseline in Hematology Parameter: Hemoglobin
Description: Blood samples were collected for the analysis of hematology parameter: hemoglobin. Baseline value was the latest pre-dose (Day -1) assessment with a non-missing value, including those from unscheduled visits. Change from Baseline is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day -1) and at 72 hours at each Treatment Period
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Placebo | GSK2982772 60 mg | GSK2982772 120 mg | GSK2982772 240 mg
Number analyzed (Participants) | 12 | 12 | 12 | 12
Grams per liter | 2.4 (6.01) | 4.6 (5.74) | -1.4 (5.57) | -0.4 (8.65)

10. Primary Outcome: Change From Baseline in Hematology Parameter: Erythrocyte Mean Corpuscular Hemoglobin (MCH)
Description: Blood samples were collected for the analysis of hematology parameter: erythrocyte MCH. Baseline value was the latest pre-dose (Day -1) assessment with a non-missing value, including those from unscheduled visits. Change from Baseline is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day -1) and at 72 hours at each Treatment Period
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Picograms
Arm/Group | Placebo | GSK2982772 60 mg | GSK2982772 120 mg | GSK2982772 240 mg
Number analyzed (Participants) | 12 | 12 | 12 | 12
Picograms | 0.12 (0.269) | 0.17 (0.299) | 0.10 (0.234) | 0.15 (0.261)

11. Primary Outcome: Change From Baseline in Hematology Parameter: Erythrocyte Mean Corpuscular Volume (MCV)
Description: Blood samples were collected for the analysis of hematology parameter: erythrocyte MCV. Baseline value was the latest pre-dose (Day -1) assessment with a non-missing value, including those from unscheduled visits. Change from Baseline is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day -1) and at 72 hours at each Treatment Period
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Femtoliters
Arm/Group | Placebo | GSK2982772 60 mg | GSK2982772 120 mg | GSK2982772 240 mg
Number analyzed (Participants) | 12 | 12 | 12 | 12
Femtoliters | -0.4 (0.90) | -0.7 (0.89) | -0.2 (0.39) | -0.4 (0.90)

12. Primary Outcome: Change From Baseline in Hematology Parameter: Erythrocytes
Description: Blood samples were collected for the analysis of hematology parameter: erythrocytes. Baseline value was the latest pre-dose (Day -1) assessment with a non-missing value, including those from unscheduled visits. Change from Baseline is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day -1) and at 72 hours at each Treatment Period
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | Placebo | GSK2982772 60 mg | GSK2982772 120 mg | GSK2982772 240 mg
Number analyzed (Participants) | 12 | 12 | 12 | 12
10^12 cells per liter | 0.058 (0.2387) | 0.126 (0.1583) | -0.059 (0.1624) | -0.035 (0.2731)

13. Primary Outcome: Change From Baseline in Hematology Parameter: Reticulocytes/Erythrocytes
Description: Blood samples were collected for the analysis of hematology parameter: percentage reticulocytes. Baseline value was the latest pre-dose (Day -1) assessment with a non-missing value, including those from unscheduled visits. Change from Baseline is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day -1) and at 72 hours at each Treatment Period
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Ratio of Reticulocytes to Erythrocytes
Arm/Group | Placebo | GSK2982772 60 mg | GSK2982772 120 mg | GSK2982772 240 mg
Number analyzed (Participants) | 12 | 12 | 12 | 12
Ratio of Reticulocytes to Erythrocytes | 0.0002 (0.00221) | 0.0001 (0.00188) | -0.0008 (0.00242) | -0.0003 (0.00201)

14. Primary Outcome: Change From Baseline in Hematology Parameters: Platelets and Leukocytes of TID Doses for One Day of GSK2982772
Description: Blood samples were collected for the analysis of hematology parameters including platelet count and leukocytes. Baseline value was the latest pre-dose (Day -1) assessment with a non-missing value, including those from unscheduled visits. Change from Baseline is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day -1) and at 72 hours at each Treatment Period
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | Placebo | GSK2982772 60 mg | GSK2982772 120 mg | GSK2982772 240 mg
Number analyzed (Participants) | 12 | 12 | 12 | 12
10^9 cells per liter
  Platelets | -1.8 (21.35) | 2.5 (26.12) | -12.8 (23.03) | -6.4 (18.59)
  Leukocytes | -0.43 (0.927) | -0.05 (0.992) | -0.42 (1.214) | -0.62 (0.860)

15. Primary Outcome: Change From Baseline in Hematology Parameters of TID Doses for One Day of GSK2982772
Description: Blood samples were collected for the analysis of hematology parameters including neutrophils/leukocytes, lymphocytes/leukocytes, monocytes/leukocytes, eosinophils/leukocytes and basophils/leukocytes. Baseline value was the latest pre-dose (Day -1) assessment with a non-missing value, including those from unscheduled visits. Change from Baseline is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day -1) and at 72 hours at each Treatment Period
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Percentage of cells in leukocytes
Arm/Group | Placebo | GSK2982772 60 mg | GSK2982772 120 mg | GSK2982772 240 mg
Number analyzed (Participants) | 12 | 12 | 12 | 12
Percentage of cells in leukocytes
  Neutrophils/Leukocytes | 0.04 (4.656) | -0.55 (4.356) | -0.75 (5.841) | -1.57 (8.363)
  Monocytes/Leukocytes | -1.13 (1.598) | -0.24 (1.019) | -0.01 (1.176) | -0.48 (1.532)
  Lymphocytes/Leukocytes | 1.29 (4.206) | 1.02 (4.329) | 1.49 (4.847) | 2.29 (8.349)
  Eosinophils/Leukocytes | -0.18 (0.666) | -0.22 (1.335) | -0.66 (1.377) | -0.27 (0.537)
  Basophils/Leukocytes | -0.02 (0.180) | -0.01 (0.090) | -0.08 (0.129) | 0.02 (0.134)

16. Primary Outcome: Change From Baseline in Urine Potential of Hydrogen (pH)
Description: Urine samples were collected for analysis of urine pH. pH is calculated on a scale of 0 to 14, values on the scale refer to the degree of alkalinity or acidity. A pH of 7 is neutral. A pH of less than 7 is acidic and a pH of greater than 7 is basic. Normal urine has a slightly acidic pH (5.0-6.0). Baseline value was the latest pre-dose (Day -1) assessment with a non-missing value, including those from unscheduled visits. Change from Baseline is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day -1) and at 72 hours at each Treatment Period
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Placebo | GSK2982772 60 mg | GSK2982772 120 mg | GSK2982772 240 mg
Number analyzed (Participants) | 12 | 12 | 12 | 12
pH | 0.13 (0.569) | 0.42 (0.515) | 0.42 (0.515) | -0.17 (0.537)

17. Primary Outcome: Change From Baseline in Urine Specific Gravity
Description: Urine samples were collected for analysis of urine specific gravity. Urine specific gravity is a measure of the concentration of solutes in the urine and provides information on the kidney's ability to concentrate urine. The concentration of the excreted molecules determines the urine's specific gravity. The urinary specific gravity measurement is a routine part of urinalysis. Baseline value was the latest pre-dose (Day -1) assessment with a non-missing value, including those from unscheduled visits. Change from Baseline is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day -1) and at 72 hours at each Treatment Period
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Ratio of urine density to water density
Arm/Group | Placebo | GSK2982772 60 mg | GSK2982772 120 mg | GSK2982772 240 mg
Number analyzed (Participants) | 12 | 12 | 12 | 12
Ratio of urine density to water density | 0.0093 (0.00702) | 0.0042 (0.00780) | 0.0068 (0.00631) | 0.0036 (0.00825)

18. Primary Outcome: Number of Participants With Abnormal Urinalysis Results by Dipstick Method
Description: Urine samples were collected to assess urine bilirubin, urine glucose, urine ketones, urine occult blood, urine protein and urine urobilinogen by dipstick test. The dipstick test gives results in a semi-quantitative manner, and results for urinalysis parameter of urine bilirubin, urine occult blood, urine glucose, urine ketones, urine protein and urine urobilinogen can be read as negative (-) and trace (+-) indicating proportional concentrations in the urine sample.
Time Frame: At 72 hours of each Treatment Period
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK2982772 60 mg | GSK2982772 120 mg | GSK2982772 240 mg
Number analyzed (Participants) | 12 | 12 | 12 | 12
Participants
  Bilirubin, 72 hours, negative | 12 | 12 | 12 | 12
  Glucose, 72 hours, negative | 12 | 12 | 12 | 12
  Ketones, 72 hours, negative | 12 | 12 | 12 | 12
  Occult Blood, 72 hours, negative | 12 | 12 | 12 | 12
  Protein, 72 hours, negative | 12 | 12 | 12 | 12
  Urobilinogen, 72 hours, trace | 12 | 12 | 12 | 12

19. Primary Outcome: Change From Baseline in Electrocardiogram (ECG) Finding: Mean Heart Rate
Description: Full 12-lead ECGs were recorded in participant using an automated ECG machine. Baseline value was the latest pre-dose (Day -1) assessment with a non-missing value, including those from unscheduled visits. Change from Baseline is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day -1) and at 2, 7, 14, 24, 48 and 72 hours at each Treatment Period
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Placebo | GSK2982772 60 mg | GSK2982772 120 mg | GSK2982772 240 mg
Number analyzed (Participants) | 12 | 12 | 12 | 12
Beats per minute
  2 hours | 3.1 (5.20) | 2.9 (4.54) | 0.6 (3.78) | 2.0 (5.86)
  7 hours | 10.7 (5.21) | 9.6 (4.72) | 9.0 (5.53) | 10.8 (7.79)
  14 hours | 6.9 (3.18) | 7.3 (4.20) | 7.7 (5.35) | 8.3 (4.18)
  24 hours | 3.0 (4.31) | 2.3 (4.03) | 2.1 (6.79) | 1.8 (4.82)
  48 hours | 0.6 (3.99) | 3.7 (3.31) | 1.3 (6.96) | 2.3 (7.62)
  72 hours | 6.2 (5.57) | 5.9 (3.20) | 3.7 (6.05) | 8.3 (5.87)

20. Primary Outcome: Change From Baseline in ECG Findings of TID Doses for One Day of GSK2982772
Description: Full 12-lead ECGs were recorded in participants using an automated ECG machine and measured PR, QRS, QT and QTcF intervals. Baseline value was the latest pre-dose (Day -1) assessment with a non-missing value, including those from unscheduled visits. Change from Baseline is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day -1) and at 2, 7, 14, 24, 48 and 72 hours at each Treatment Period
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Placebo | GSK2982772 60 mg | GSK2982772 120 mg | GSK2982772 240 mg
Number analyzed (Participants) | 12 | 12 | 12 | 12
Milliseconds
  PR interval, 2 hours | -3.7 (8.22) | -2.3 (7.62) | 0.5 (8.36) | -4.0 (7.48)
  PR interval, 7 hours | -9.5 (13.70) | -8.3 (7.95) | -3.8 (11.77) | -7.0 (10.04)
  PR interval, 14 hours | -7.5 (9.95) | -0.8 (11.92) | -0.2 (10.77) | -4.2 (11.00)
  PR interval, 24 hours | 1.2 (7.26) | -0.2 (8.07) | 1.7 (9.18) | 1.5 (13.32)
  PR interval, 48 hours | 2.0 (13.75) | 1.0 (9.89) | 2.8 (11.98) | 3.7 (7.33)
  PR interval, 72 hours | -0.2 (15.92) | 1.2 (8.20) | 2.0 (13.43) | 4.8 (13.47)
  QRS duration, 2 hours | -2.3 (6.60) | -2.7 (7.69) | -2.2 (7.16) | 0.3 (4.89)
  QRS duration, 7 hours | 0.7 (6.95) | -0.5 (4.52) | -0.5 (6.39) | 1.7 (4.33)
  QRS duration, 14 hours | 3.5 (8.40) | 0.8 (1.59) | 0.3 (5.52) | 1.5 (7.34)
  QRS duration, 24 hours | 1.3 (5.14) | 0.7 (3.34) | -1.3 (7.74) | 0.7 (5.99)
  QRS duration, 48 hours | 1.0 (6.12) | -1.3 (5.28) | -0.2 (10.50) | -2.5 (5.13)
  QRS duration, 72 hours | 1.0 (4.47) | 0.2 (5.62) | 1.0 (8.33) | 0.3 (4.96)
  QT interval, 2 hours | -8.0 (13.56) | -3.2 (22.94) | -9.8 (20.69) | -4.7 (17.53)
  QT interval, 7 hours | -22.7 (18.79) | -29.7 (15.06) | -22.2 (22.33) | -31.3 (24.10)
  QT interval, 14 hours | -20.5 (17.35) | -21.3 (17.55) | -20.0 (20.47) | -23.5 (20.91)
  QT interval, 24 hours | -8.3 (13.59) | 0.7 (14.95) | -13.5 (16.65) | -6.7 (13.84)
  QT interval, 48 hours | -3.3 (9.55) | -7.3 (10.39) | -15.2 (20.85) | -15.7 (17.24)
  QT interval, 72 hours | -18.0 (17.20) | -11.8 (13.42) | -14.7 (20.44) | -23.3 (12.69)
  QTcF interval, 2 hours | -0.1 (16.40) | 4.0 (19.41) | -7.1 (18.60) | 0.6 (17.64)
  QTcF interval, 7 hours | 2.1 (15.02) | -6.7 (15.07) | -1.4 (16.59) | -7.2 (14.83)
  QTcF interval, 14 hours | -3.6 (16.50) | -3.8 (12.75) | -1.4 (13.94) | -4.8 (15.60)
  QTcF interval, 24 hours | -0.5 (14.44) | 7.8 (15.82) | -7.8 (19.60) | -1.8 (9.04)
  QTcF interval, 48 hours | -1.9 (13.55) | 1.9 (7.18) | -11.3 (12.20) | -10.0 (16.31)
  QTcF interval, 72 hours | -2.9 (12.92) | 2.6 (11.37) | -4.8 (13.30) | -4.5 (12.26)

21. Primary Outcome: Number of Participants With Abnormal Not Clinically Significant Cardiac Telemetry
Description: Continuous cardiac telemetry was performed and number of participants with abnormal clinically significant and not clinically significant values are presented.
Time Frame: Up to 24 hours at each Treatment Period
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK2982772 60 mg | GSK2982772 120 mg | GSK2982772 240 mg
Number analyzed (Participants) | 12 | 12 | 12 | 12
Participants
  Abnormal-not clinically significant | 1 | 0 | 0 | 0
  Abnormal-clinically significant | 0 | 0 | 0 | 0

22. Primary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: Blood pressure of participants were measured at indicated time points in supine position after 5 minutes rest. Baseline value was the latest pre-dose (Day -1) assessment with a non-missing value, including those from unscheduled visits. Change from Baseline is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day -1) and at 2, 7, 14, 24, 48 and 72 hours at each treatment period
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Placebo | GSK2982772 60 mg | GSK2982772 120 mg | GSK2982772 240 mg
Number analyzed (Participants) | 12 | 12 | 12 | 12
Millimeters of mercury
  DBP, 2 hours | 0.2 (5.13) | -2.5 (7.22) | -1.9 (5.73) | -2.2 (8.09)
  DBP, 7 hours | -7.3 (6.75) | -7.0 (8.12) | -8.2 (8.33) | -5.9 (8.75)
  DBP, 14 hours | -4.4 (5.16) | -5.3 (8.29) | -6.9 (5.88) | -4.3 (8.88)
  DBP, 24 hours | -2.2 (6.15) | 0.3 (6.41) | -4.0 (5.24) | -2.4 (10.21)
  DBP, 48 hours | -1.3 (6.88) | 1.3 (5.83) | -0.3 (4.69) | 0.5 (9.30)
  DBP, 72 hours | -0.2 (5.25) | 0.3 (6.66) | -0.1 (7.18) | 2.8 (10.84)
  SBP, 2 hours | 1.3 (6.85) | 0.4 (7.55) | 2.4 (4.10) | 0.6 (5.30)
  SBP, 7 hours | -0.3 (8.99) | 2.5 (6.65) | -0.7 (8.15) | 1.3 (6.09)
  SBP, 14 hours | 3.3 (5.76) | 1.0 (6.06) | 9.0 (11.24) | 5.6 (11.12)
  SBP, 24 hours | 0.3 (4.70) | 0.1 (5.55) | 1.4 (6.07) | 2.9 (5.93)
  SBP, 48 hours | 0.8 (6.05) | -0.3 (6.24) | 1.2 (4.26) | -1.1 (5.52)
  SBP, 72 hours | 1.9 (9.23) | 2.3 (8.57) | 3.8 (7.57) | 4.5 (5.04)

23. Primary Outcome: Change From Baseline in Pulse Rate of TID Doses for One Day of GSK2982772
Description: Pulse rate of participants were measured at indicated time points in supine position after 5 minutes rest. Baseline value was the latest pre-dose (Day -1) assessment with a non-missing value, including those from unscheduled visits. Change from Baseline is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day -1) and at 2, 7, 14, 24, 48 and 72 hours at each Treatment Period
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Placebo | GSK2982772 60 mg | GSK2982772 120 mg | GSK2982772 240 mg
Number analyzed (Participants) | 12 | 12 | 12 | 12
Beats per minute
  2 hours | 0.9 (5.35) | 1.7 (4.19) | 0.4 (4.10) | 0.8 (3.81)
  7 hours | 6.9 (4.17) | 9.4 (5.60) | 8.9 (5.92) | 10.4 (6.75)
  14 hours | 3.3 (3.50) | 5.3 (3.58) | 5.5 (4.44) | 8.3 (4.50)
  24 hours | -0.9 (4.74) | 1.0 (3.64) | 1.1 (2.75) | 3.3 (4.11)
  48 hours | -1.7 (3.98) | 1.5 (3.37) | 1.3 (4.97) | 4.3 (5.45)
  72 hours | -0.4 (6.57) | 5.0 (3.79) | 2.2 (4.91) | 6.0 (5.48)

24. Primary Outcome: Change From Baseline in Body Temperature of TID Doses for One Day of GSK2982772
Description: Temperature of participants were measured at indicated time points in supine position after 5 minutes rest. Baseline value was the latest pre-dose (Day -1) assessment with a non-missing value, including those from unscheduled visits. Change from Baseline is calculated as the value at the post-dose visit minus the Baseline value.
Time Frame: Baseline (Day -1) and at 2, 7, 14, 24, 48 and 72 hours at each Treatment Period
Population: Safety Population.
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | Placebo | GSK2982772 60 mg | GSK2982772 120 mg | GSK2982772 240 mg
Number analyzed (Participants) | 12 | 12 | 12 | 12
Degrees Celsius
  2 hours | 0.22 (0.204) | 0.32 (0.199) | 0.12 (0.241) | 0.18 (0.276)
  7 hours | 0.47 (0.274) | 0.51 (0.231) | 0.43 (0.261) | 0.48 (0.366)
  14 hours | 0.39 (0.264) | 0.48 (0.191) | 0.40 (0.388) | 0.65 (0.258)
  24 hours | 0.07 (0.223) | -0.05 (0.239) | 0.08 (0.237) | 0.08 (0.286)
  48 hours | 0.06 (0.297) | -0.07 (0.235) | -0.08 (0.222) | 0.12 (0.292)
  72 hours | 0.09 (0.257) | 0.00 (0.191) | 0.09 (0.284) | 0.24 (0.271)

25. Primary Outcome: Number of Participants With Abnormal Neurological Examinations of TID Doses for One Day of GSK2982772
Description: Neurological examinations including: mental status, gait, balance, coordination, cranial nerves, motor power, reflexes, and sensory system (light touch and pain) were assessed in participants specified time points.
Time Frame: Baseline (Day -1) and at 2, 7, 14, 24, 48 and 72 hours at each Treatment Period
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK2982772 60 mg | GSK2982772 120 mg | GSK2982772 240 mg
Number analyzed (Participants) | 12 | 12 | 12 | 12
Participants | 0 | 0 | 0 | 0

26. Secondary Outcome: Area Under the Plasma Drug Concentration Versus Time Curve Over 24 Hours (AUC[0-24]) and AUC Over Each Dose Interval of TID Doses for One Day of GSK2982772
Description: Blood samples were collected from participants at indicated time points and analyzed for AUC (0-24) and AUC over each dose: AUC(0-7), AUC (7-14) and AUC (14-24) after the administration of TID doses of GSK2982772. Pharmacokinetic analysis was conducted using standard non-compartmental methods. All participants in the safety population for whom a pharmacokinetic sample has been obtained and analyzed was included in the pharmacokinetic population.
Time Frame: Pre-dose, 20 and 40 minutes, 1, 1.5, 2, 3, 5, 7 hours, 7 hours 20 minutes, 7 hours 40 minutes, 8, 8.5, 9, 10, 12, 14 hours, 14 hours 20 minutes, 14 hours 40 minutes, 15, 15.5, 16, 17, 19, 22 and 24 hours post-dose at each Treatment Period
Population: Pharmacokinetic Population. Only those participants with data available at the specified data points were analyzed (represented by n=X in the category titles).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | GSK2982772 60 mg | GSK2982772 120 mg | GSK2982772 240 mg
Number analyzed (Participants) | 12 | 12 | 12
Hours*microgram per milliliter
  AUC (0-24), n=12, 12, 12 | 13.153 (22.4) | 25.779 (17.7) | 54.960 (19.0)
  AUC (0-7), TID dose 1, n=10, 10, 7: number analyzed (Participants) | 10 | 10 | 7
  AUC (0-7), TID dose 1, n=10, 10, 7 | 3.804 (22.4) | 6.553 (22.6) | 10.854 (26.6)
  AUC (7-14), TID dose 2, n=10, 6, 8: number analyzed (Participants) | 10 | 6 | 8
  AUC (7-14), TID dose 2, n=10, 6, 8 | 4.684 (18.7) | 9.200 (18.6) | 20.875 (20.5)
  AUC (14-24), TID dose 3, n=12, 12, 12 | 4.919 (24.9) | 10.105 (20.8) | 23.602 (16.8)

27. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) and Observed Trough Drug Plasma Concentrations Following Each TID Doses for One Day of GSK2982772
Description: Blood samples were collected from participants at indicated time points and analyzed for Cmax and observed trough drug plasma concentrations: C0, C7, C14 and C24 after the administration of TID doses of GSK2982772.
Time Frame: Pre-dose,20 and 40 minutes, 1, 1.5, 2, 3, 5, 7 hours,7 hours 20 minutes,7 hours 40 minutes,8, 8.5, 9, 10, 12, 14 hours,14 hours 20 minutes,14 hours40 minutes, 15, 15.5, 16, 17, 19, 22, 24, 28, 32, 36, 48, 60 and 72 hours post-dose at each Treatment Period
Population: as for outcome 26
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter
Arm/Group | GSK2982772 60 mg | GSK2982772 120 mg | GSK2982772 240 mg
Number analyzed (Participants) | 12 | 12 | 12
Micrograms per milliliter
  Cmax, TID dose 1, n=12, 12, 12 | 1.187 (16.2) | 2.003 (27.7) | 3.038 (27.5)
  Cmax, TID dose 2, n=12, 12, 12 | 1.322 (34.2) | 2.727 (21.2) | 5.516 (21.1)
  Cmax, TID dose 3, n=12, 12, 12 | 1.076 (32.9) | 2.378 (17.8) | 5.120 (13.2)
  C0, TID dose 1, n=0, 0, 0: number analyzed (Participants) | 0 | 0 | 0
  C7, TID dose 1, n=12, 12, 12 | 0.149 (55.3) | 0.344 (41.5) | 0.878 (54.7)
  C14, TID dose 2, n=12, 12, 12 | 0.175 (44.0) | 0.439 (44.6) | 0.999 (26.5)
  C24, TID dose 3, n=12, 12, 12 | 0.107 (44.7) | 0.229 (53.3) | 0.543 (47.6)

28. Secondary Outcome: Terminal Half Life (t1/2) After the Third TID Dose for One Day of GSK2982772
Description: Blood samples were collected from participants at indicated time points and t1/2 was analyzed after the administration of third TID dose of GSK2982772.
Time Frame: as for outcome 27
Population: Pharmacokinetic Population. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | GSK2982772 60 mg | GSK2982772 120 mg | GSK2982772 240 mg
Number analyzed (Participants) | 12 | 12 | 11
Hours | 5.883 (52.5) | 7.206 (31.9) | 6.624 (51.8)

29. Secondary Outcome: Time to Maximum Observed Plasma Drug Concentration (Tmax) of Each TID Doses for One Day of GSK2982772
Description: Blood samples were collected from participants at indicated time points and Tmax was analyzed after the administration of TID doses of GSK2982772.
Time Frame: as for outcome 27
Population: Pharmacokinetic Population.
Measure: Median (Full Range); unit: Hours
Arm/Group | GSK2982772 60 mg | GSK2982772 120 mg | GSK2982772 240 mg
Number analyzed (Participants) | 12 | 12 | 12
Hours
  TID dose 1 | 2.000 [1.00 to 3.00] | 1.750 [1.00 to 3.00] | 2.000 [1.50 to 5.00]
  TID dose 2 | 1.750 [1.00 to 3.00] | 2.500 [1.50 to 5.00] | 2.000 [1.50 to 3.00]
  TID dose 3 | 2.500 [0.67 to 5.00] | 3.000 [1.00 to 5.00] | 3.000 [2.00 to 3.00]

ADVERSE EVENTS:
Time Frame: Non-serious AEs and SAEs were collected from the start of the treatment up to 39 days
Description: Non-serious AEs and SAEs were collected for Safety population
Arm/Group | Placebo | GSK2982772 60 mg | GSK2982772 120 mg | GSK2982772 240 mg
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 1/12 | 0/12 | 0/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=12) | GSK2982772 60 mg (N=12) | GSK2982772 120 mg (N=12) | GSK2982772 240 mg (N=12)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-06-27): https://cdn.clinicaltrials.gov/large-docs/13/NCT03590613/Prot_001.pdf
  • Statistical Analysis Plan (2018-07-11): https://cdn.clinicaltrials.gov/large-docs/13/NCT03590613/SAP_000.pdf